CLINICAL TRIAL: NCT00327483
Title: Web Based Renal Transplant Patient Medication Education
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Educational/Counseling/Training
Other Study IDs: R01HS015038-03 (AHRQ)
Record Dates: First submitted 2006-05-16; First posted 2006-05-18 (Estimated); Last update posted 2006-05-18 (Estimated); Status verified 2006-05

CONDITIONS: Renal Transplant Recipients
Keywords: Transplant; Medication error; Patient Safety; Information technology

INTERVENTIONS:
Behavioral: Internet based education software

SUMMARY:
Information technology will be brought directly to renal transplant recipients to help them learn about the large number of medications they are required to take on a life long basis, in order to prevent errors and improve safety.

DETAILED DESCRIPTION:
Transplant recipients are particularly vulnerable to medication errors because of the large number of chronic drugs needed to prevent rejection and treat comorbidities. Compliance failures directly compromise patient safety through acute immunologic events and premature graft loss. For society, the loss of invested fiscal and organic (organs) resources is catastrophic. As the unique constant in the chain of people who provide, modify and consume prescription medications, health information technology should be focused on empowering the patient to prevent medication errors. Our principal clinical hypothesis is that HIT can be proven to improve patient safety by minimizing medication errors. Specific aims address the creation of new knowledge and evidence ( in a renal transplant population) of benefits of widely applicable HIT tools. Web enabled education of two groups, new (<6 months) and established (> 6 months), kidney transplant recipients is proposed.

ELIGIBILITY:
Inclusion Criteria:age > 18 or capable of managing own medications

-

Exclusion Criteria:Education level below 10th grade

-

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 250
Dates: Start 2005-07; Study Completion 2006-04

PRIMARY OUTCOMES:
Medication errors

SECONDARY OUTCOMES:
Serum creatinine
Rejection episodes
Rehospitalizations
Graft loss

CONTACTS AND LOCATIONS:
Overall Officials: Amy L Friedman, MD, Principal Investigator — Yale University
Locations (1):
- Yale New Haven Hospital, New Haven, Connecticut, United States